CLINICAL TRIAL: NCT05339347
Title: A Sham-controlled Crossover Study Using Photoneuromodulation to Treatment the Negative Symptoms of Schizophrenia.
Brief Title: Schizophrenia Treatment With Photoneuromodulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leandro Valiengo, Medical Assistance, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4.545.487
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Photoneuromodulation; Neuromodulation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: For the sham, the tip has LED light similar to the real one, but without generating the light field. The treatments will be administered in two sessions (active/sham) with a Light-Aid (Bright Photomedicine, SP, Brazil), continuous wave, 300 LEDs, wavelength of 850 nm). The irradiation parameters created will be based on the skin phototype according to the Fitzpatrick Scale.
  The tip will be positioned in the prefrontal cortex (corresponding to F3 and F4 according to the 10-20 EEG system). This arrangement is commonly known as 'Bifrontal'. In each application, power densities between 45-50 mW/cm², frequency of 10 Hz, and total time of 10 to 15 minutes per session will be used. The tip used has a size equivalent to 70cm² each side.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We have two identical devices (a and b), that are equal in all aspects, but one of them is sham (does not product infrared (IR) light). As IR light is invisible for human eyes, neither the applicant of the procedure neither the participant will know if it is active or sham. All the participants had a code after randomization that does the allocation to sham or active. The machine (a or b) was chosen for an external researcher that has no contact with the team of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: Active Photoneuromodulation (Active Comparator): Active stimulation with light fields as described in the intervention
  Interventions: Device: Photoneuromodulation
- Sham Comparator: Sham Photoneuromodulation (Sham Comparator): The blinding will be done with sham light, which consists of fields that do not reproduce light, but which have the same size and thickness as the true one.
  Interventions: Device: Photoneuromodulation

INTERVENTIONS:
Device: Photoneuromodulation — Treatments were administered daily for a period of 2 weeks (10 sessions) with a Light-Aid (Bright Photomedicine, SP, Brazil), continuous wave, 300 LED wavelength 850 nm) or with a placebo probe of the same appearance and display. The irradiation parameters created will be based on the disease, pain intensity and skin phototype. Each session has from 10 to 15 min, depending on skin phototype

SUMMARY:
Abstract: Randomized clinical trial that aims to see the efficacy of photoneuromodulation for the treatment of negative symptoms of schizophrenia in patients refractory to transcranial direct current stimulation. In this group of 30 refractory volunteers, magnetic resonance spectroscopy will be performed before and after photoneuromodulation in a cross-over design.

Objectives: Effectiveness of photoneuromodulation in patients with schizophrenia. . Analysis of glutamate, Gaba and lactate in spectroscopy before and after stimulation (secondary) Sample: 30 volunteers with negative symptoms of schizophrenia refractory to treatment.

Method: clinical trial, cross-over randomized, double-blind, sham-controlled. PANSS negative symptoms subscale evaluation before and after the 10 photoneuromodulation sessions. Participants who are in the active group after the 10 photoneuromodulation sessions will go to the sham group and vice versa. They will perform magnetic resonance spectroscopy before the beginning, after the 10 sessions and again after the inversion of the groups (3 resonances per volunteer). The study will be a cross-over: half of participants will start at sham group and the other half at active group and invert groups after 10th day of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 55 years
* Diagnosis of schizophrenia according to DSM-IV criteria and confirmed by the SCID (Structured Clinical Interview for DSMIV), which will be applied by a psychiatrist, will be included.
* Minimum score of 20 points in the sum of negative PANSS
* Stable antipsychotic medications
* There is a need for at least one trial with at least one antipsychotic in adequate dose and time to enter the study.

Exclusion Criteria:

* Unstable or uncontrolled clinical diseases,
* Psychiatric comorbidities,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Changes in Subcale of PANSS | Weeks 0, 2 and 4
  Continuos measure (score changes)

SECONDARY OUTCOMES:
Changes in PANSS | Time Frame: Weeks 0, 1, 2, 3, 4, 6, 12]
  Continuous measure (score changes).
Changes in WHOQOL | Time Frame: Weeks 0, 1, 2, 3, 4, 6, 12]
  Continuous measure (score changes).
Changes in Brief Negative Symptom Scale (BNSS) | Time Frame: Weeks 0, 1, 2, 3, 4, 6, 12]
  Continuous measure (score changes).
Changes in Calgary | Time Frame: Weeks 0, 1, 2, 3, 4, 6, 12]
  Continuous measure (score changes).
Changes in SOFAS | Time Frame: Weeks 0,1, 2, 3, 4, 6, 12]
  Continuous measure (score changes).
Changes in SANS | Time Frame: Weeks 0, 1, 2, 3, 4, 6, 12]
  Continuous measure (score changes).
Changes in parameters of spectroscopy (lactate, glutamate, glicine and GABA) | Time Frame: Weeks 0, 2, 4]
  Continuous measure (score changes).

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Valiengo, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No